CLINICAL TRIAL: NCT01960153
Title: Phosphodiesterase Type 5 Inhibition With Tadalafil Changes Outcomes in Heart Failure: Extent of Renal Damage (PITCH-ER)
Brief Title: Phosphodiesterase Type 5 Inhibition With Tadalafil Changes Outcomes in Heart Failure: Extent of Renal Damage
Acronym: PITCH-ER
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Award was ended by NIH for parent study
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Carelon Research (Other)
Responsible Party: Principal Investigator, Ravi Thadhani, Chief, Division of Nephrology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2013P001412; R01HL119155-01A1 (NIH)
Record Dates: First submitted 2013-10-08; First posted 2013-10-10 (Estimated); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Heart Failure; Pulmonary Hypertension
Keywords: Heart failure; Pulmonary hypertension; tadalafil; Phosphodiesterase Type 5 Inhibition
MeSH Terms: conditions — Heart Failure; Hypertension, Pulmonary | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tadalafil (Experimental): Tadalafil is supplied in 20 mg tablets. Subjects will take 20 mg (one tablet) once per day and will be titrated to 40 mg (two tablets once per day) after one week. Subjects are on study drug for the duration of the trial.
  Interventions: Drug: Tadalafil
- Placebo (Placebo Comparator): Placebo of tadalafil. Subjects will take one tablet once per day and will be titrated to two tablets once per day after one week. Subjects are on study drug for the duration of the trial.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tadalafil — Tadalafil tablets, 20 mg to 40 mg per day x 48 weeks
  Other Names: Adcirca
  Arms: Tadalafil
Drug: Placebo — Placebo of tadalafil. Subjects will take one tablet once per day and will be titrated to two tablets once per day after one week. Subjects are on study drug for the duration of the trial.
  Arms: Placebo

SUMMARY:
PITCH-ER is an ancillary study of PITCH-HF (NCT01910389). The goal of the PITCH-ER ancillary study is to evaluate the rate of decline in renal function and frequency of development of acute kidney injury (AKI) in patients enrolled in PITCH-HF (who have heart failure and pulmonary hypertension) treated with chronic tadalafil treatment compared to placebo.

DETAILED DESCRIPTION:
The National Heart, Lung, and Blood Institute (NHLBI)-funded parent study (PITCH-HF) is the first well-controlled, randomized, large-scale trial studying the effect of tadalafil, an FDA-approved selective phosphodiesterase type 5 inhibitor (PDE5i), on cardiovascular and heart failure-related deaths and hospitalizations in patients with heart failure and secondary pulmonary hypertension.

Both chronic kidney disease (CKD), as reflected by albuminuria and reduced estimated glomerular filtration rate (eGFR) and acute kidney injury (AKI) significantly contribute to morbidity and mortality in the population of patients who will be enrolled in PITCH-HF. Therapies that alter the course of renal disease in patients with heart failure are lacking. The biology of treatment with PDE5i strongly suggests a potential protective effect of these agents on renal function.

This ancillary PITCH-ER study leverages the PITCH-HF infrastructure and randomization, adding only longitudinal collection of subjects' urine samples to 5 timepoints throughout the study. With these urine samples collected, PITCH-ER will address 2 major patient-oriented questions:

1. Does chronic tadalafil treatment slow the rate of GFR decline and/or modify the development/progression of albuminuria vs placebo? To answer this question, longitudinal measures of eGFR utilizing state-of-the-art equations that incorporate serum creatinine and cystatin C and spot urine albumin-to-creatinine ratios (UACR) will be measured.
2. Does PDE5i treatment reduce AKI frequency and/or the magnitude of urinary biomarker changes reflecting subclinical renal injury vs placebo? An AKI adjudication committee will monitor the incidence of AKI events and their severity using the Kidney Disease Improving Global Outcomes (KDIGO) consensus criteria. Subclinical renal injury will be detected using validated urinary biomarkers: neutrophil gelatinase-associated lipocalin (NGAL) and kidney injury marker 1 (KIM-1).

Since 30% of the overall PITCH-HF population will likely have diabetes (which amplifies the risk for renal injury in HF patients), PITCH-ER will repeat analyses in the population stratified by baseline diabetes status as secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* All subjects eligible for enrollment into the PITCH-HF parent trial are eligible to enroll in this ancillary study (Refer to PITCH-HF NCT01910389 for specific eligibility criteria)

Exclusion Criteria:

* Subjects who are not eligible for enrollment into the PITCH-HF parent trial may not enroll in this ancillary study (Refer to PITCH-HF NCT01910389 for specific eligibility criteria)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2017-12 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Change in renal function | Baseline to 48 months
  Between-group differences in changes from baseline in: (1a) eGFR using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation and (1b) spot urine albumin-to-creatinine ratio (UACR)
Incidence of acute kidney injury (AKI) events (clinical and subclinical) | Baseline to 48 months
  Impact of treatment on (2a) incidence of AKI events (adjudicated) based on new Kidney Disease Improving Global Outcomes criteria; and (2b) changes from baseline in the urine biomarkers of subclinical kidney injury: Neutrophil Gelatinase-Associated Lipocalin (NGAL) and Kidney Injury Marker 1 (KIM-1).

SECONDARY OUTCOMES:
Changes in renal function stratified by diabetes/no diabetes | Baseline to 48 months
  As for the primary outcome, measurements will be eGFR and UACR
Incidence of AKI events stratified by diabetes/no diabetes | Baseline to 48 months
  As for the primary outcome, AKI events will be adjudicated and N-GAL and KIM-1 will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Ravi I Thadhani, MD, MPH, Principal Investigator — Massachusetts General Hospital; Ishir Bhan, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- See also: PITCH-HF Parent Study — http://clinicaltrials.gov/ct2/show/record/NCT01910389